CLINICAL TRIAL: NCT06281184
Title: Long-term Effects of Methotrexate in Adults With Erosive Hand Osteoarthritis: A 30-month Follow-up of Former MERINO Participants (MERINO:2).
Brief Title: A 30-month Follow-up of MERINO Participants to Evaluate Long-term Effects of Methotrexate in Erosive Hand OA.
Acronym: MERINO:2
Status: Enrolling by invitation | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DIA2024.1; 715758 (Registry Identifier: Regional committee for medical and health research ethics)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hand Osteoarthritis; Erosive Osteoarthritis
Keywords: Erosive hand osteoarthritis
MeSH Terms: interventions — Methotrexate; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- MTX -- MTX: MERINO trial: randomized to methotrexate (MTX) MERINO:2 study: continues with MTX
  Interventions: Drug: Methotrexate
- MTX -- Treatment as usual: MERINO trial: randomized to methotrexate (MTX) MERINO:2 study: continues without MTX
  Interventions: Other: Treatment as usual
- Placebo -- MTX: MERINO trial: randomized to placebo MERINO:2 study: continues with MTX
  Interventions: Drug: Methotrexate
- Placebo -- Treatment as usual: MERINO trial: randomized to placebo MERINO:2 study: continues without MTX
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 5-25 mg x 1 per week, combined with folic acid 1mg daily.
  Groups: MTX -- MTX; Placebo -- MTX
Other: Treatment as usual — No specific treatment after MERINO-trial
  Groups: MTX -- Treatment as usual; Placebo -- Treatment as usual

SUMMARY:
In response to the high prevalence of synovitis in hand osteoarthritis (OA) and its association with pain, there's a compelling rationale for investigating the efficacy of MTX in managing inflammatory erosive hand OA. Recent guidelines highlight the need for large, well-designed trials to assess the effectiveness of MTX. A recent trial (METHODS study) showed promising pain reduction with MTX, but due to pandemic-related protocol changes, the duration of the study was limited to six months. The ongoing MERINO trial randomizes participants to MTX or placebo for one year. After completing the MERINO trial, several participants asked for MTX open label. In the subsequent MERINO:2 study, participants completing the trial will be invited to a structured follow-up after one year, including electronic questionnaires and hand radiographs, providing valuable long-term data on the effects of MTX in hand OA. Together, these trials aim to fill gaps in understanding the long-term impact of MTX in hand OA, particularly on structural progression.

DETAILED DESCRIPTION:
The primary aim is to demonstrate the superiority of Methotrexate (MTX) over no treatment in slowing radiographic progression over 24 months in individuals with erosive hand osteoarthritis (OA).

OA is a leading cause of disability and affecting millions worldwide, with a significant impact on knee, hip, and hand joints. Despite its high prevalence and symptomatic burden, effective disease-modifying treatments remain elusive, with current options limited to pain management and joint replacement.

MTX, recognized for its disease-modifying effects in systemic inflammatory joint diseases, offers promising potential in OA treatment, with previous trials indicating its anti-inflammatory properties and potential for joint damage reduction. In the ongoing MERINO trial, 153 participants are randomly assigned to either MTX or a placebo. Following completion of the trial, several participants have expressed interest in MTX treatment, which is sometimes used off-label for erosive hand OA patients experiencing unmanageable pain and inflammation. As a result, some MERINO trial participants will receive MTX treatment.

In the MERINO:2 study, we will conduct a structured follow-up one year post-MERINO trial completion, incorporating hand radiographs and pain questionnaires. This endeavor will furnish invaluable insights into the long-term effects of MTX treatment in erosive hand OA, a gap in current knowledge, particularly regarding structural progression. This will provide valuable data on long-term effects of MTX treatment in erosive hand OA, which is not currently described in the literature, especially on structural progression.

ELIGIBILITY:
Eligible participants are those enrolled in the MERINO-trial (EudraCT number 2019-004641-33, Clincaltrials.gov number NCT04579848, REK ID 2020/187524, CTIS number 2023-510523-30-00).

Inclusion Criteria:

* Finger joint pain 40-80 on 0-100 visual analog scale (VAS) with insufficient pain relief from, inability to tolerate or contra-indications to oral paracetamol and/or NSAIDs, and hand symptoms (pain, aching, or stiffness) on most days the previous 6 weeks before randomization.
* Hand OA according to the American College of Rheumatology (ACR) criteria, at least 1 distal (DIP) or proximal interphalangeal (PIP) joint of the 2nd-5th finger with radiographic pre-erosive (J-phase) or erosive disease (E-phase) according to the Verbruggen-Veys anatomical phase system, and at least two DIP/PIP joints with power Doppler signal of at least grade 1 or grey-scale synovitis of at least grade 2 on ultrasound.

Exclusion Criteria:

* Contraindications to methotrexate:

  * Abnormal renal function, defined as serum creatinine >142 µmol/L in women and >168 µmol/L in men, or a glomeruli filtration rate (GFR) <40 mL/min/1.73 m2.
  * Abnormal liver function, defined as transaminases above the upper normal limit, active or previous hepatitis B or C infection, or known cirrhosis
  * Lung fibrosis (maximum 6 months old x-ray), active infection, or reduced hematopoiesis (i.e. anemia, leukopenia and/or thrombocytopenia).
  * Planned pregnancy within 18 months after screening (men/women), and pregnancy, breastfeeding, or insufficient anti-conception therapy for female fertile participants. Contraception should be maintained during treatment and until the end of systemic exposure, i.e. 3 months after methotrexate discontinuation. Sufficient anti-conception therapy consists of intra-uterine device (coil) or hormonal anti-conception (birth control pills, implant, intra-uterine system, dermal patch, vaginal ring, or injections).
  * Alcohol or other drug abuse in the last year.
  * Intolerance to lactose.
* Chronic inflammatory rheumatic diseases (such as rheumatoid arthritis and psoriatic arthritis or gout), active inflammatory bowel disease, or positive rheumatoid factor or anti-CCP antibodies.
* Other severe co-morbidities such as hemochromatosis, fibromyalgia, psoriasis, blood dyscrasias, and coagulation disorders, history of malignancy (except successfully treated squamous or basal cell skin carcinoma), uncontrolled diabetes mellitus, severe hypertension, unstable ischemic heart disease, severe heart failure, severe pulmonary disease, severe and/or opportunistic infections and/or chronic infections, active tuberculosis, positive human immunodeficiency virus (HIV) status, recent stroke, bone marrow hypoplasia, or demyelinating diseases of the central nervous system.
* Other likely causes of hand symptoms: thoracic outlet syndrome, carpal tunnel disease, diabetic cheiropathy, injury in finger joints previous 6 months, or palmar tenosynovitis/trigger finger.
* Oral or intra-muscular steroids in the previous month
* Intra-articular treatments or aspirations of any kind of any joint in the hands 3 months before inclusion
* Analgesics or NSAIDs, unless stable dosage for ≥1 month.
* Symptomatic slow-acting drugs for OA (SYSADOA), unless stable dose for ≥3 months and require stable dose throughout the study.
* Disease-modifying osteoarthritis drugs (DMOADs) previous three months.
* Scheduled hand surgery during study participation.
* Planning to start other treatments for hand OA in the study participation period.
* Not able to adhere to the study visit schedule and protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are those enrolled in the MERINO-trial (EudraCT number 2019-004641-33, Clincaltrials.gov number NCT04579848, REK ID 2020/187524, CTIS number 2023-510523-30-00).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of MTX on radiographic progression of erosive hand OA. | 18 months
  Effect of MTX on radiographic progression of erosive hand OA according to Verbruggen-Veys anatomical atlas score at 12 months

SECONDARY OUTCOMES:
Effect of MTX on pain, function and life quality | 18 months
  • Finger joint pain previous 48 hours (VAS) at 18 months • Thumb base joint pain previous 48 hours (VAS) at 18 months • Pain most painful finger joint previous 48 hours (VAS) at 18 months • AUSCAN pain and function subscales at 18 months • OMERACT-OARSI responder criteria at 18 months • Patient-reported disease activity previous 48 hours (VAS) at 18 months • EQ-5D at 18 months
Effect of MTX on radiographic progression of hand OA. | 18 months
  • KL grades • OARSI atlas (osteophytes, joint space narrowing, erosions)

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT06281184/Prot_000.pdf
  • Informed Consent Form: English version (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT06281184/ICF_001.pdf
  • Informed Consent Form: Norwegian version (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT06281184/ICF_002.pdf